CLINICAL TRIAL: NCT06366776
Title: Emulated Clinical Trial of the Influence of Corrected Low 25-OH Vitamin D Levels on Healthcare Costs and Healthcare Utilization
Brief Title: Emulated Study of Vitamin D Correction Vs Non-Correction
Status: Active, not recruiting | Type: Observational
Sponsor: The Cooper Health System (Other)
Collaborators: Won Sook Chung Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23-278
Record Dates: First submitted 2024-03-12; First posted 2024-04-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-04

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; healthcare cost; healthcare utilization; hospitalization; emergency room visit; intensive care unit admission; emulated trial; target trial; real world data; combined comorbidity; multimorbidity; propensity score
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Treatment Group: Any patient with a 25-OH vitamin D level(s) always lower than 40 ng/ml (low level) with subsequent level(s) in the 40 ng/ml to 100 ng/ml range. The 40 ng/ml to 100 ng/ml range is maintained for three years.
- Control Group A: Any patient with a 25-OH vitamin D level always lower than 40 ng/ml with maintenance of that lower than 40 ng/ml level for 3 years.
- Control Group B: Any patient who has an uninterrupted 25-OH vitamin D level greater than or equal 40 ng/ml and less than or equal to 100 ng/ml (sufficient level) for a continuous 3-year period. Prior to the 3-year period there were no levels lower than 40ng/ml or higher than 100 ng/ml.

SUMMARY:
* This is a single-site retrospective electronic chart review of Cooper Health System Inpatients and Outpatients from 2008 through 2023 aged eighteen years or older. This review is designed as an emulation of a randomized clinical trial with a nonrandomized database.
* The primary objectives are to compare healthcare costs and healthcare utilization between subjects who have corrected low vitamin D levels and those without corrected low vitamin D levels.

DETAILED DESCRIPTION:
* The purpose of the study is to characterize healthcare costs and healthcare utilization in subjects with corrected low (<40 ng/ml) 25-OH vitamin D levels compared to subjects with uncorrected low 25-OH vitamin D levels during a three-year period.
* The primary objective of this study is to determine whether ten healthcare costs are lower and ten healthcare utilization parameters occur less frequently in patients with corrected low vitamin D levels compared to patients with uncorrected low vitamin D levels in Cooper outpatients and inpatients.

The costs are:

1. total billed costs for any reason;
2. total billed costs for hospitalizations;
3. total billed costs for ICU admissions;
4. total billed costs for emergency room visits;
5. total billed costs for all other outpatient services;
6. total billed costs for urgent care visits;
7. total billed costs for primary care physician (PCP) services;
8. total billed costs for nurse practitioner (NP) services;
9. total billed costs for all other professional services;
10. total billed costs for medical pharmacy services and products.

The parameters are:

1. number of hospitalizations for any reason;
2. number of ICU admissions for any reason;
3. number of emergency room visits for any reason;
4. all other outpatient services for any reason;
5. number of urgent care visits for any reason;
6. number of primary care physician visits for any reason;
7. number of nurse practitioner visits for any reason;
8. all other professional services for any reason;
9. number of medical pharmacy services for any reason;
10. number of free-standing prescriptions for any reason.

    * The secondary objective is to determine the effect of sufficient vitamin D levels (≥ 40 ng/ml) in subjects not requiring a prior correction on the ten healthcare costs parameters and the ten healthcare utilization parameters listed in the primary objective above.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with at least one 25-OH vitamin D test result. Patients with one test result will remain in the limited dataset for potential future research.
* Any patient with a 25-OH vitamin D level(s) always lower than 40 ng/ml (low level) with subsequent level(s) in the 40 ng/ml to 100 ng/ml range. The 40 ng/ml to 100 ng/ml range is maintained for three years. This corrected group is labeled as the Treatment Group.
* Any patient with a 25-OH vitamin D level always lower than 40 ng/ml with maintenance of that lower than 40 ng/ml level for 3 years. This uncorrected group is labeled as Control Group A.
* Any patient who has an uninterrupted 25-OH vitamin D level greater than or equal 40 ng/ml and less than or equal to 100 ng/ml (sufficient level) for a continuous 3-year period. Prior to the 3-year period there were no levels lower than 40ng/ml or higher than 100 ng/ml. This vitamin D3 sufficient group is labeled as Control Group B.

Exclusion Criteria:

* Any patient with only one 25-OH vitamin D3 test result or any patient who cannot be included in the Treatment Group, Control Group A, or Control Group B is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators anticipate reviewing records from thousands of patients in order to identify enough patients that meet the eligibility criteria. Investigators will enroll at a minimum 3,000 patients in the Treatment Group and at a minimum 3,000 patients in Control Group A regarding the primary objective. In regard to the secondary objective, the investigators will enroll as many as available for Control Group B.
Sampling Method: Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Ten healthcare costs parameters among the corrected Treatment Group and the uncorrected Control Group A. | 3 year observation period
  The ten healthcare costs parameters: total billed costs for any reason; costs for hospitalizations; costs for ICU admissions; costs for emergency room visits; costs for all other outpatient services; costs for urgent care visits; costs for primary care physician (PCP) services; costs for nurse practitioner (NP) services; costs for all other professional services; and costs for medical pharmacy services and products among Treatment Group and Control Group A..
Ten healthcare utilization parameters among the corrected Treatment Group and the uncorrected Control Group A. | 3 year observation period
  The ten healthcare utilization parameters: number of hospitalizations; number of ICU admissions; number of emergency room visits; all other outpatient services; number of urgent care visits; number of primary care physician services; number of nurse practitioner services; all other professional services; number of medical pharmacy services or products; and number of free-standing prescriptions among Treatment Group and Control Group A.

SECONDARY OUTCOMES:
Ten healthcare costs parameters among patients with sufficient vitamin D levels (Control Group B). | 3 year observation period
  The secondary outcomes are the ten healthcare costs parameters listed in the primary outcomes above relating to patients with sufficient vitamin D levels who did not require a prior correction (Control Group B).
Ten healthcare utilization parameters among patients with sufficient vitamin D levels (Control Group B). | 3 year observation period
  The secondary outcomes are the ten healthcare utilization parameters listed in the primary outcomes above relating to patients with sufficient vitamin D levels who did not require a prior correction (Control Group B).

CONTACTS AND LOCATIONS:
Overall Officials: Ludmil Mitrev, MD, Principal Investigator — Cooper Health System
Locations (1):
- Cooper Health System, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No